CLINICAL TRIAL: NCT00506558
Title: The CSM Trial: A Multicenter Study Comparing Ventral to Dorsal Surgery for Cervical Spondylotic Myelopathy
Acronym: CSM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Greenwich Hospital (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH-CSM-382; GH-CSM-382
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Cervical Spondylotic Myelopathy
Keywords: cervical spondylotic myelopathy; degenerative cervical spondylosis; spinal fusion
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Ventral Decompression and Instrumented Fusion
  Interventions: Procedure: Ventral Surgical Decompression with Instrumented Fusion
- B (Active Comparator): Dorsal Decompression with or without fusion
  Interventions: Procedure: Dorsal Decompression With or Without Fusion

INTERVENTIONS:
Procedure: Ventral Surgical Decompression with Instrumented Fusion — Multi-level discectomy or Corpectomy are performed at surgeon's discretion. After decompression an instrumented fusion is performed.
  Arms: A
Procedure: Dorsal Decompression With or Without Fusion — Dorsal decompressive laminectomy, laminoplasty, or laminectomy with lateral mass instrumented fusion
  Arms: B

SUMMARY:
The purpose of the study is to determine the optimal surgical approach (ventral versus dorsal) for patients with multi-level cervical spondylotic myelopathy (CSM). There are no established guidelines for the management of patients with CSM, which slowly causes spinal cord injury in afflicted patients.

This study aims to test the hypothesis that ventral surgery (decompressing the spinal cord from the front of the neck) and dorsal surgery (decompressing the spinal cord from the back of the neck) might differ in their overall outcome or major complication rate.

DETAILED DESCRIPTION:
A. Purpose To determine the optimal surgical approach (ventral versus dorsal) for patients with multi-level cervical spondylotic myelopathy (CSM).

B. Background There are no established guidelines for the management of patients with CSM. It is estimated that up to 30 percent of patients have an unsatisfactory outcome after surgery for CSM. It remains uncertain how dorsal and ventral approaches differ in their success rates and in their complication rates. This study aims to test the hypothesis that ventral and dorsal surgical approaches differ in their outcomes or major complication rates. A secondary hypothesis is that fusion might improve outcome by reducing repetitive shear injury to the spinal cord.

C. Specific Location of Study

This is a multi-center trial. Subjects will be entered into the study from 9 separate centers. At this site, subjects will be recruited from the office of Dr. Zoher Ghogawala. All subjects at this site will undergo surgery at Greenwich Hospital.

D. Probable Duration of Project

Subjects will be recruited into the study for one year. All subjects will be followed for 1 year.

E. Research Plan

1. Prospective, non-randomized multicenter trial. Approximately 100-200 patients would be recruited over one year with follow-up at one year.
2. Subjects (aged 40-85 years) with spinal cord compression (2 or more levels) from degenerative cervical spondylosis with clinical myelopathy will be treated with either ventral decompression/fusion or dorsal decompression with or without fusion.
3. Subjects with cervical kyphosis > 5˚, a segmental kyphotic deformity defined as 3 or more disc-osteophytes that extend dorsal to a line drawn from the dorsal caudal point of C2 to the dorsal caudal point of C7, ossification of the posterior longitudinal ligament (OPLL), or developmental spinal canal narrowing (12mm) would be excluded from the study.
4. Functional outcomes will be determined using well-known quantitative scales (SF-36, Oswestry Neck, mJOA, Nurick, and EuroQol-5D). These instruments will be administered pre-op, 3 months, 6 months, and 1 year post-op.
5. Two independent neuroradiologists will review the initial films to confirm eligibility and review post-operative films (3 months, 6 months, and 1 year) to determine radiographic decompression and fusion as well as any complications.
6. An independent study coordinator will collect data at 30 days and at 1 year to document any complications or re-operations.

F. Data and Safety Monitoring Plan

1. All serious unexpected adverse events (e.g. death within 30 days of operation) will be reported to the IRB within 24 hours. Any appropriate funding agencies or regulatory agencies would be notified as well.
2. Any serious anticipated adverse event (e.g. wound infection, pulmonary embolus) will be reported to the IRB whenever their magnitude or frequency exceeds expectations.
3. All other adverse events (including loss of privacy, significant economic harm) will be reported to the IRB on an annual basis or at the time that re-approval is sought. Any adverse event judged unlikely or unrelated to the study will also be included in an annual report for the IRB.

G. Statistical Considerations

1. Specific data variables being collected for the study.

   The data collection sheets will be submitted along with this protocol. There will be several data sheets as follows: 1) Spine surgeon's data sheet, 2) 30-day and 6-month morbidity data sheet, 3)1-year morbidity data sheet, 4) SF-36 questionnaires (pre-op, 3 months, 6 months, 1 year), 5) Oswestry Neck Disability Index questionnaires (pre-op, 3 months, 6 months, 1 year), 6)mJOA, (pre-op, 3 months, 6 months, 1 year), 7) Nurick questionnaire (pre-op, 3 months, 6 months, 1 year), 8)EuroQol-5D (pre-op, 3 months, 6 months, 1 year), 9)Radiology Review (pre-op, 3 months, 6 months, 1 year, 2 years).
2. Study endpoints.

   Patients will be followed for 1 year. The primary endpoints will be the SF-36 physical component summary score (PCS) and the Oswestry Neck Disability Index. Secondary endpoints will include the Nurick, mJOA, and EuroQol-5D scores as well as the observed complication rates. Radiographic fusion, instability, and deformity will also be secondary outcomes.
3. Statistical Methods.

   Analysis will focus on the physical component summary (PCS) of the SF-36, the Oswestry Neck Disability index, and the major complication rate. The t-test will be used to compare the groups for continuous variables such as the SF-36 PCS and the Oswestry Neck Disability Index. The Chi-square test will be used to compare the group's complication rates. Multiple regression techniques will be applied to control for potential confounders including age, medical condition, number of stenotic levels, degree of lordosis or kyphosis, etc.
4. Power Analysis.

The data generated from the SF-36 or the Oswestry Neck Disability Index will be used to calculate sample size for a future randomized controlled trial (RCT) comparing ventral to dorsal surgery. If no significant differences are identified in these primary outcomes measures, then a sample size calculation will be done using any differences in major complication rates.

ELIGIBILITY:
Inclusion Criteria:

* degenerative cervical spondylotic myelopathy (2 or more levels of spinal cord compression)

Exclusion Criteria:

* C2-C7 kyphosis>5˚ (measured on lateral cervical spine image in extension)
* Segmental kyphotic deformity defined as 3 or more levels of disc-osteophyte extend dorsal to a line drawn from the dorsal caudal point of C2 to the dorsal caudal point of C7.
* Ossification of posterior longitudinal ligament (OPLL)
* Developmental narrow canal (<12 mm-canal diameter measured on lateral plain cervical spine film)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Oswestry Neck Disability Index, mJOA, major complication rate | 1 year

SECONDARY OUTCOMES:
SF-36 physical component summary (PCS), EuroQol-5D | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Ghogawala, MD, FACS, Study Director — Greenwich Hospital - Yale Universtiy School of Medicine; Edward C. Benzel, MD, Principal Investigator — The Cleveland Clinic; Robert Heary, MD, Principal Investigator — University of Medicine and Dentistry of New Jersey; Ronald Apfelbaum, Principal Investigator — University of Utah; Jean-Valery Coumans, MD, Principal Investigator — Massachusetts General Hospital; Subu N Magge, MD, Principal Investigator — Lahey Clinic
Locations (7):
- United States (7):
  - Danbury Hospital, Danbury, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Medicine and Dentistry - New Jersey, Newark, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Utah HSC, Salt Lake City, Utah

REFERENCES:
- [Background] Fessler RG, Steck JC, Giovanini MA. Anterior cervical corpectomy for cervical spondylotic myelopathy. Neurosurgery. 1998 Aug;43(2):257-65; discussion 265-7. doi: 10.1097/00006123-199808000-00044. PMID 9696078
- [Background] Edwards CC 2nd, Heller JG, Murakami H. Corpectomy versus laminoplasty for multilevel cervical myelopathy: an independent matched-cohort analysis. Spine (Phila Pa 1976). 2002 Jun 1;27(11):1168-75. doi: 10.1097/00007632-200206010-00007. PMID 12045513
- [Result] Ghogawala Z, Coumans JV, Benzel EC, Stabile LM, Barker FG 2nd. Ventral versus dorsal decompression for cervical spondylotic myelopathy: surgeons' assessment of eligibility for randomization in a proposed randomized controlled trial: results of a survey of the Cervical Spine Research Society. Spine (Phila Pa 1976). 2007 Feb 15;32(4):429-36. doi: 10.1097/01.brs.0000255068.94058.8a. PMID 17304133